CLINICAL TRIAL: NCT00719758
Title: TRK-100STP Pharmacokinetic Study in Healthy Volunteers - Evaluation of Pharmacokinetic Interaction Between TRK-100STP and Kremezin
Brief Title: Drug-Drug Interaction Study of TRK-100STP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Toray Industries, Inc (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 533-CL-005
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: TRK-100STP,; beraprost sodium,; Careload LA; AST-120; Spherical carbon adsorbent; Drug-drug interaction
MeSH Terms: interventions — beraprost; AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cross-over study
  Interventions: Drug: TRK-100STP (BERASUS LA); Drug: AST-120 (Kremezin®)

INTERVENTIONS:
Drug: TRK-100STP (BERASUS LA) — oral
  Other Names: beraprost; Careload LA; BERASUS LA
Drug: AST-120 (Kremezin®) — oral
  Other Names: Kremezin®; sopherical carbon adsorbent

SUMMARY:
The purpose of this study is to evaluate the effect of AST-120 on the PK of TRK-100STP, and to evaluate the safety and tolerability of TRK-100STP alone or in combination with AST-120

DETAILED DESCRIPTION:
Non-blinded, randomized and crossover study to evaluate pharmacokinetic interaction between TRK-100STP and AST-120 in different administration condition. Nonelderly adult volunteers will receive TRK-100STP with or without AS-T120 after meal. Safety parameters will concurrently be measured.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Body Mass Index (BMI) of ≥17.6 to ≤26.4 kg/m2 and weight of ≥50 to ≤80 kg

Exclusion Criteria:

* Clinical abnormal physical findings, including BP, pulse rate, ECG and laboratory assessments
* Receives any investigational medicine within 120 days before screening
* Recent blood donor

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | 1 day

SECONDARY OUTCOMES:
Safety parameters (vital signs, ECG, laboratory tests) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan